CLINICAL TRIAL: NCT00062387
Title: A Phase II Study Of Perifosine In Patients With Recurrent Or Metastatic Head And Neck Cancer
Brief Title: Perifosine in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02538; UCCRC-12198A; NCI-5938; CDR0000304740 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2004-10

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — perifosine

ARMS (1):
- Arm I (Experimental): Patients receive oral perifosine 4 times daily on days 1 and 2 and once daily on days 3-28 during course 1. Patients receive oral perifosine once daily on days 1-28 for all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: perifosine

INTERVENTIONS:
Drug: perifosine

SUMMARY:
Phase II trial to study the effectiveness of perifosine in treating patients who have recurrent or metastatic head and neck cancer. Drugs used in chemotherapy such as perifosine use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the antitumor activity of perifosine in patients with recurrent or metastatic squamous cell head and neck cancer.

II. Determine the time to progression and overall survival of patients treated with this drug.

III. Determine the toxicity of this drug in these patients. IV. Determine the pharmacodynamics of this drug in these patients. V. Assess the usefulness of biomarkers in predicting response and other outcome parameters in patients treated with this drug.

VI. Assess the quality of life of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral perifosine 4 times daily on days 1 and 2 and once daily on days 3-28 during course 1. Patients receive oral perifosine once daily on days 1-28 for all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, weekly during the first month, every 28 days after the first month, and then at study withdrawal.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 22-46 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell cancer of the head and neck

  * Metastatic or recurrent disease
  * Not amenable to surgery or radiotherapy
* Unidimensionally measurable disease

  * At least 1 lesion at least 20 mm by conventional techniques OR at least 10 mm by CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to perifosine
* No ongoing or active infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 1 prior biologic/targeted regimen for recurrent or metastatic disease

Chemotherapy

* No more than 1 prior adjuvant or neoadjuvant chemotherapy and/or concurrent chemoradiotherapy regimen
* No more than 1 prior chemotherapy regimen for recurrent or metastatic disease
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Radiotherapy

* At least 4 weeks since prior radiotherapy

Other

* Recovered from prior therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (12):
- United States (12):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Argiris A, Cohen E, Karrison T, Esparaz B, Mauer A, Ansari R, Wong S, Lu Y, Pins M, Dancey J, Vokes E. A phase II trial of perifosine, an oral alkylphospholipid, in recurrent or metastatic head and neck cancer. Cancer Biol Ther. 2006 Jul;5(7):766-70. doi: 10.4161/cbt.5.7.2874. Epub 2006 Jul 2. PMID 16760642